CLINICAL TRIAL: NCT01800383
Title: Cerebral GABA and Fear Conditioning in PTSD
Status: Completed | Type: Observational
Sponsor: Isabelle Rosso (Other)
Collaborators: Mclean Hospital (Other)
Responsible Party: Sponsor-Investigator, Isabelle Rosso, Director, Anxiety and Traumatic Stress Disorders Laboratory, Mclean Hospital
Organization: Mclean Hospital (Other)
Other Study IDs: MH096987-01A1
Record Dates: First submitted 2013-02-14; First posted 2013-02-27 (Estimated); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: posttraumatic stress disorder; fear conditioning; proton magnetic resonance spectroscopy; GABA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Control: No Axis I psychiatric disorder and no trauma exposure
- Trauma-Exposed Normal Control: History of trauma exposure and subthreshold PTSD symptoms.
- PTSD: Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis of PTSD as determined by the Structured Clinical Interview for DSM-IV-Text Revised

SUMMARY:
Posttraumatic stress disorder (PTSD) is a common and debilitating neuropsychiatric disorder in which an acute fear response to a traumatic event does not abate. This failure to recover from trauma is thought to be due at least in part to a deficit in learning not to fear situations and stimuli previously associated with the trauma (i.e., specifically due to a failure of extinction recall). Pavlovian fear conditioning can be simulated and measured experimentally in humans using a 2-day fear conditioning paradigm developed by our group, wherein conditioning and extinction learning phases are conducted on Day 1, and extinction recall is tested on Day 2.

Recent functional magnetic resonance imaging (fMRI) evidence indicates that PTSD is associated with hyper-responsivity of the insular cortex and hyporesponsivity of the ventromedial prefrontal cortex (VMPFC) during exposure to fear-inducing stimuli, consistent with altered excitability of brain regions mediating fear conditioning and extinction. As the brain's principal inhibitory neurotransmitter, GABA exerts a prominent role in modulating neuronal excitability. Interestingly, there are reports that adjunctive treatment with GABA-enhancing antiepileptics is efficacious in PTSD. There is also evidence, albeit inconsistent, that lower serum GABA levels predict a more chronic course of the illness. However, it is unclear whether serum levels accurately reflect brain GABA, which may contribute to inconsistency of serum findings. Moreover, it is possible that GABA alterations may vary in their presence, nature and significance across brain regions implicated in PTSD. The proposed study will examine the relationship of PTSD symptoms and behavioral fear conditioning deficits with regional brain gamma-aminobutyric acid (GABA) using proton magnetic resonance spectroscopy (1H-MRS).

We have the following aims and hypotheses:

1. To determine whether GABA alterations are associated with the categorical diagnosis of PTSD and not merely exposure to trauma. It is hypothesized that PTSD will be associated with higher GABA in VMPFC and lower GABA in the right insula.
2. To determine whether GABA levels are significantly associated with dimensional measures of PTSD symptom severity and individual symptom dimensions. It is predicted that higher GABA in the VMPFC and lower GABA in the right anterior insula will be associated with greater total symptom severity.
3. To determine whether GABA in VMPFC and right anterior insula are significantly associated with measures of extinction recall failure and anxiety sensitivity in PTSD. It is hypothesized that VMPFC GABA will be positively correlated with skin conductance response to a conditioned stimulus that had previously been extinguished and insula GABA will be negatively correlated with anxiety sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* 20-50 years of age
* right-handed
* DSM-IV diagnosis consistent with group assignment
* groups to be matched for age, sex, education, race/ethnicity
* ability to provide written informed consent
* groups to be matched on proportion of female subjects in follicular/luteal menstrual phases.

Exclusion Criteria:

* Medical condition that would confound results
* history of seizures or head trauma with loss of consciousness
* exposure to psychotropic medications within 4 weeks of study (8 weeks for fluoxetine)
* metal implants, claustrophobia or other Magnetic Resonance Imaging (MRI) exclusions
* positive urine toxicology or human chorionic gonadotropin (HCG) status on scan day
* history of psychotic disorder, bipolar disorder, eating disorder, mental retardation, or pervasive developmental disorder; history of meeting full criteria for non-PTSD anxiety disorder.
* PTSD and trauma subjects will be matched in terms of comorbid depressive disorder, not to exceed 50%. Trauma-exposed subjects will have a history of trauma exposure and will not meet criteria for PTSD. Non-traumatized healthy subjects will have no history of Axis I psychiatric disorder and no trauma exposure.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be between the ages of 20 and 50 years. These will include 31 subjects meeting DSM-IV criteria for PTSD, 31 trauma-exposed healthy subjects, and 31 healthy comparison (HC) subjects without any trauma exposure.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Regional brain gamma-aminobutyric acid (GABA) levels in the ventromedial prefrontal cortex (VMPFC), right anterior insula, and right posterior temporal cortex | Measured on the day of the MRI scan
  Single voxel 3T H-MRS cortex using a MEGAPRESS sequence will be used to detect and quantify GABA in these brain regions.
Regional brain glutamate metabolism in the ventromedial prefrontal cortex (VMPFC), right anterior insula, and right posterior temporal cortex | Measured on the day of the MRI scan
  Single voxel 3T H-MRS cortex using a 2DJPRESS sequence at 3T will be used to detect and quantify glutamate and glutamine in these brain regions.
Regional brain neuronal integrity in the ventromedial prefrontal cortex (VMPFC), right anterior insula, and right posterior temporal cortex | Measured on the day of the MRI scan
  Single voxel 3T H-MRS cortex using a 2DJPRESS sequence at 3T will be used to detect and quantify N-acetyl aspartate in these brain regions.

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States